CLINICAL TRIAL: NCT03350841
Title: Evaluation of Post-operative Pain Following Platelet Rich Plasma (PRP) Revascularization Versus Conventional Endodontic Treatment of Non-vital Mature Mandibular Molars With Chronic Peri-apical Periodontitis
Brief Title: Pain After PRP Revascularization and Endodontic Treatment of Non-vital Mandibular Molars With Apical Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yassmin Elsayed Ahmed, Assisstant lecturer-endodontic department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-11-27
Record Dates: First submitted 2017-11-16; First posted 2017-11-22 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revascularization (Experimental): platelet rich plasma injected in the canals
  Interventions: Procedure: Platelet rich plasma PRP
- root canal treatment (Active Comparator): endodontic treatment obturated with gutta percha
  Interventions: Procedure: root canal treatment

INTERVENTIONS:
Procedure: Platelet rich plasma PRP — blood sample is collected to prepare platelet rich plasma injected in the canal
  Arms: Revascularization
Procedure: root canal treatment — conventional root canal treatment and obturation with guttapercha
  Arms: root canal treatment

SUMMARY:
randomized clinical trial which Evaluate thr Post-operative Pain Following Platelet Rich Plasma (PRP) Revascularization versus Conventional Endodontic Treatment of Non-vital Mature Mandibular Molars with Chronic Peri-apical Periodontitis

DETAILED DESCRIPTION:
it will be done in 2 visits where in the firist visit, i will finish cleaning and shaping of the canals and inject double antibiotic paste as intracanal medication.

in the second visit, removal of intracanal medication then obturaton of the canals in the control group. while in the intervention group,over instrumentation of the canals beyond the working length using k-file size 20-35 to establish bleeding in the canals.then blood sample is collected for PRP preparation then injected into the canal.the patient will record post operative pain 6,12,24,48 hours then 3,4,5 days later.then they will do CBCT at 6, 12 months after the treatment to assess peri-apical healing

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients, between 18-40 years
* Patients with necrotic pulp in mandibular molar permanent teeth with closed apex

Exclusion Criteria:

* Illiterate patient
* Patients with systemic diseases
* Pregnant women
* Patients that have allergy to ciprofloxacin or metronidazole
* Teeth that:

  * Have vertical root fracture, coronal perforation, and calcification.
  * re-treatment cases
  * Non restorable
* Patients that have T.M.J. disorder

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative Pain | 5 days
  postoperative pain evaluated using NRS scale It is a numerical rating scale from 0-10 with 0 representing no pain and 10 representing worst pain

SECONDARY OUTCOMES:
healing | 12 months
  healing of periapical tissue evaluated radiographically

CONTACTS AND LOCATIONS:
Locations (1):
- Yassmin Elsayed Ahmed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided